CLINICAL TRIAL: NCT04101396
Title: 4 Versus 7 Points Self-monitoring Blood Glucose in Gestational Diabetes on Diet Modification-A Randomised Control Trial
Brief Title: 4 vs 7 Points Blood Glucose Monitoring in Gestational Diabetes on Dietary Modification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Rahana Abd Rahman, Principal Investigator, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FF-2019-351
Record Dates: First submitted 2019-09-17; First posted 2019-09-24 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: diet modification, 4 and 7 points monitoring
MeSH Terms: interventions — Diet, Diabetic

STUDY DESIGN:
Intervention Model Description: All women with gestational diabetes are randomised to 4 or 7 points of self monitoring blood glucose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 points blood glucose monitoring (Other): 4 points of self monitoring blood glucose which comprises of fasting, 1 hour post breakfast, 1 hour post lunch and 1 hour post dinner
  Interventions: Dietary Supplement: diabetic diet
- 7 points blood glucose monitoring (Other): 7 points of self monitoring blood glucose which comprises of fasting,1 hour post breakfast, 1 hour pre and post lunch, 1 hour pre and post dinner, pre bed at 10 pm
  Interventions: Dietary Supplement: diabetic diet

INTERVENTIONS:
Dietary Supplement: diabetic diet — Patients with gestational diabetes will be seen by the dietitian to be taught diet modification

SUMMARY:
This study aims to compare between 4 and 7 points blood glucose monitoring in women with gestational diabetes on diet modification.

DETAILED DESCRIPTION:
All women with gestational diabetes on diet modification will be recruited and randomised to 4 versus 7 points self monitoring blood glucose. They will be followed up 4 weekly and the pregnancy outcomes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years old
* Pregnant women with gestational diabetes mellitus on diet modification
* Confirmed gestational diabetes mellitus using National Institute for Health and Care Excellence guideline by 75g oral glucose tolerance test after 14 weeks
* Gestational age at recruitment 20-34 week

Exclusion Criteria:

* bad obstetrics history.
* Women with underlying medical disorders such as hypertension, autoimmune diseases on steroids
* fetal anomaly.
* Women planning to deliver in other centres
* Women who refuse to participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Pregnancy outcome of participants | From date of randomisation up to 40 weeks gestation
  Mean gestational age at delivery in weeks
Pregnancy outcome of participants | From date of randomisation up to 40 weeks gestation and participants are diagnosed in established labour
  Rate of spontaneous or induced labour in percentage
Pregnancy outcome of participants | From date of randomisation up to 40 weeks gestation when the participants had given birth to the newborn
  Rate of vaginal, instrumental or caesarean delivery in percentage
Pregnancy outcome of participants | From date of randomisation up to 40 weeks gestation during progress of labour up to 24 hours post delivery
  Rate of intrapartum complications such as postpartum haemorrhage, shoulder dystocia and third or fourth degree tear in percentage
Pregnancy outcome of participants | At the point of birth of the neonate
  Mean neonatal birth weight in kilogram
Pregnancy outcome of participants | At the point of birth of the neonate
  Rate of neonates born with Apgar score at five minutes of less than 7 in percentage
Pregnancy outcome of participants | At the point of birth of the neonate
  Rate of neonatal intensive care unit admission in percentage
Pregnancy outcome of participants | From date of randomisation up to 7 days after birth of the neonate
  Rate of neonatal complications such as intrauterine fetal demise, neonatal death, neonatal hypoglycaemia, neonatal jaundice, neonatal respiratory distress syndrome and neonatal sepsis in percentage
Demographic data of participants | On the date of randomisation
  Mean age of participants in years
Demographic data of participants | On the date of randomisation
  Rate of each different races such as Malay, Chinese and Indian in percentage
Demographic data of participants | On the date of randomisation
  Rate of parity such as nulliparous or multiparous in percentage
Demographic data of participants | On the date of randomisation up to 40 weeks gestation based on the first trimester weight documented in the antenatal record
  Mean prepregnancy body mass index in kg/m^2
Demographic data of participants | On the date of randomisation till 40 weeks gestation
  Mean total weight gain in kilogram
Demographic data of participants | On the date of randomisation up to 40 weeks gestation
  Rate of positive family history of diabetes mellitus in percentage
Demographic data of participants | On the date of randomisation up to 40 weeks gestation
  Rate of previous pregnancy affected by gestational diabetes mellitus in percentage
Demographic data of participants | On the date of randomisation up to 40 weeks gestation
  Rate of previous pregnancy complicated by fetal macrosomia in percentage
Clinical characteristics of participants | On the date of randomisation up to 40 weeks gestation
  Mean gestational age gestational diabetes mellitus is diagnosed in weeks
Clinical characteristics of participants | On the date of randomisation up to 40 weeks gestation
  Mean fasting glucose level from the modified glucose tolerance test in mmol/l
Clinical characteristics of participants | On the date of randomisation up to 40 weeks gestation
  Mean two hours post 75 gram glucose load from the modified glucose tolerance test in mmol/l
Clinical characteristics of participants | At the point of randomisation till 40 weeks gestation
  Rate of antenatal complications such as preeclampsia, threatened preterm labour, preterm prelabour rupture of membranes, anaemia,
Clinical characteristics of participants | At the point of randomisation till 40 weeks gestation
  Mean level of glycosylated haemoglobin in percentage
Clinical characteristics of participants | At the point of randomisation till 40 weeks gestation
  Mean level of serum fructosamine in percentage
Clinical characteristics of participants | At the point of randomisation till 40 weeks gestation
  Mean level of fasting blood glucose in self monitoring blood glucose in mmol/l
Clinical characteristics of participants | At the point of randomisation till 40 weeks gestation
  Mean level of pre-meal blood glucose in self monitoring blood glucose in mmol/l
Clinical characteristics of participants | At the point of randomisation till 40 weeks gestation
  Mean level of one hour post-meal blood glucose in self monitoring blood glucose in mmol/l

SECONDARY OUTCOMES:
Requirement of treatment in participants | From the date of randomisation up to 40 weeks gestation
  Mean gestational age that the participants are detected to require added treatment in weeks
Requirement of treatment in participants | From point of randomisation till 40 weeks gestation
  Rate of type of treatment needed such as oral hypoglycaemic agent only, combination of insulin and oral hypoglycaemic agent
Participants' compliance | From point of randomisation till 40 weeks gestation
  Rate of frequency of four weekly self blood glucose monitoring in percentage
Participants' satisfaction | From point of randomisation till 40 weeks gestation
  Rate of participants' satisfaction whether satisfied, neutral or not satisfied in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Noor Dalila Berohan, Principal Investigator — National University of Malaysia; Norasyikin Abd Wahab, Study Director — National University of Malaysia; Shuhaila Ahmad, Study Chair — National University of Malaysia
Locations (2):
- Malaysia (2):
  - Antenatal clinic, UKM Medical Centre, Cheras, Kuala Lumpur
  - National University of Malaysia, Cheras, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No
The IPD will only be shared upon request. The data that can be shared will be the blood glucose levels and pregnancy outcomes.

REFERENCES:
- [Derived] Berohan ND, Alias H, Ishak S, Mohammed Nawi A, Azman N, Sohaimi D, Kamisan Atan I, Abd Wahab N, Kalok AH, Mohamad AS, Abd Rahman R. 4 vs 7 points self-monitoring blood glucose in gestational diabetes mellitus on diet modification: randomised clinical trial in a single tertiary centre in Malaysia. Arch Gynecol Obstet. 2024 Oct;310(4):1959-1965. doi: 10.1007/s00404-024-07661-5. Epub 2024 Aug 7. PMID 39110209